CLINICAL TRIAL: NCT02381743
Title: The mCME Project:Delivering Continuing Medical Education for Community Health Workers Via SMS Text Messages
Acronym: mCME project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Christopher J. Gill, Associate Professor Global Health, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-33241
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Medical Knowledge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (No Intervention): Weekly non-medical SMS messages
- Group 2 (Experimental): Receipt of a daily SMS text message describing various aspects of clinical practice
  Interventions: Behavioral: Group 2 intervention daily SMS bullet point
- Group 3 (Experimental): Receipt of a daily SMS text message describing various aspects of clinical practice, but phrased as multiple choice question
  Interventions: Behavioral: Group 3 intervention daily SMS bullet point

INTERVENTIONS:
Behavioral: Group 2 intervention daily SMS bullet point — Group 2 subjects receive a daily SMS bullet point, summarizing a key clinical point pertinent to the CBPA's daily work.
  Other Names: non interactive model CME
  Arms: Group 2
Behavioral: Group 3 intervention daily SMS bullet point — Group 3 subjects receive a c phrased as a multiple choice question. The content mirrors that of group 2, but is presented as a question to render it interactive
  Other Names: Interactive model CME
  Arms: Group 3

SUMMARY:
Community health workers (CHWs) provide essential basic medical care to hundreds of millions of people across the globe. CHWs offer a myriad of services including community sanitation, breast feeding counseling, family planning, management of febrile children, and malaria control and prevention, to name but a few. In fact, CHWs are often the only source of primary health care available to some of the most disadvantaged populations in the world. However, to be effective, CHWs must be trained - and retrained - at regular intervals, and the costs for such trainings can be substantial. In the US, clinicians are required to stay current and maintain their competence through continuing medical education (CME). Increasingly, CME activities are delivered via internet-based, self-teaching modules. A typical example would be a set of topical readings followed by multiple-choice questions, with the answers, and CME credit, provided to the user upon satisfactory completion of the module. This content is typically delivered over the Internet. However, there is no intrinsic reason why this approach could not be adapted so that CME activities are delivered using standard cell phones via SMS text messaging. This would significantly expand professional training opportunities to a far greater range of CHWs than possible through computer/tablet/smart phone platforms, and would be particularly valuable in poorer countries with limited training budgets. In the mCME project, the investigators propose to test the effectiveness and cost effectiveness of a mobile phone-based CME delivery strategy among Vietnamese community-based physician assistants (CBPAs), a cadre of CHW mandated to provide primary health care to rural and disadvantaged populations. The investigators hypothesize that providing CME activities over a mobile platform will significantly improve their professional knowledge, and may also improve their job satisfaction and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Graduated from a CBPA training program
2. Possesses their own cell phone
3. Phone able to send/receive text messages
4. Aged 18 years or older

Exclusion Criteria:

1. Unwilling to sign informed consent
2. Lives/operates in an area without cellular coverage
3. Unwilling to be randomized
4. Unwilling to adhere to study procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Medical knowledge (Score on medical knowledge exams) | 6 months
  Score on medical knowledge exams administered at baseline and at the end of six months of the intervention

SECONDARY OUTCOMES:
Job satisfaction (Score on likert scale) | 6 months
  Score on likert scale measuring job satisfaction
Self efficacy (Score in likert scale) | 6 months
  Score in likert scale measuring self efficacy

OTHER OUTCOMES:
cost effectiveness analysis of the mCME intervention in terms of costs to increase a study test score by X % | Duration of project
  costs and cost effectiveness analysis of the mCME intervention in terms of costs to increase a study test score by X %

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gill, MD MS, Principal Investigator — Boston University

REFERENCES:
- [Derived] Larson Williams A, Hawkins A, Sabin L, Halim N, Le Ngoc B, Nguyen VH, Nguyen T, Bonawitz R, Gill C. Motivating HIV Providers in Vietnam to Learn: A Mixed-Methods Analysis of a Mobile Health Continuing Medical Education Intervention. JMIR Med Educ. 2019 Apr 18;5(1):e12058. doi: 10.2196/12058. PMID 30998220
- [Derived] Gill CJ, Le NB, Halim N, Chi CTH, Nguyen VH, Bonawitz R, Hoang PV, Nguyen HL, Huong PTT, Larson Williams A, Le NA, Sabin L. mCME project V.2.0: randomised controlled trial of a revised SMS-based continuing medical education intervention among HIV clinicians in Vietnam. BMJ Glob Health. 2018 Feb 26;3(1):e000632. doi: 10.1136/bmjgh-2017-000632. eCollection 2018. PMID 29527350
- [Derived] Gill CJ, Le Ngoc B, Halim N, Nguyen Viet H, Larson Williams A, Nguyen Van T, McNabb M, Tran Thi Ngoc L, Falconer A, An Phan Ha H, Rohr J, Hoang H, Michiel J, Nguyen Thi Thanh T, Bird L, Pham Vu H, Yeshitla M, Ha Van N, Sabin L. The mCME Project: A Randomized Controlled Trial of an SMS-Based Continuing Medical Education Intervention for Improving Medical Knowledge among Vietnamese Community Based Physicians' Assistants. PLoS One. 2016 Nov 18;11(11):e0166293. doi: 10.1371/journal.pone.0166293. eCollection 2016. PMID 27861516